CLINICAL TRIAL: NCT01071369
Title: A Randomized, Prospective, Double-Blind Controlled Evaluation of the Effectiveness of Cervical and Thoracic Interlaminar Epidural Injections in Thoracic and Cervical Disc Herniation, Discogenic Pain, and Post-Cervical Laminectomy Syndrome
Brief Title: Treatment of Chronic Thoracic and Neck and Upper Extremity Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pain Management Center of Paducah (Other)
Responsible Party: Principal Investigator, Laxmaiah Manchikanti, MD, Medical Director, Pain Management Center of Paducah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: protocol 16
Record Dates: First submitted 2008-02-14; First posted 2010-02-19 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Back Pain; Neck Pain
MeSH Terms: conditions — Back Pain; Neck Pain | interventions — Lidocaine; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomly assigned to groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Xylocaine (Active Comparator): 0.5% Xylocaine
  Interventions: Drug: Xylocaine
- Xylocaine and Celestone (Active Comparator): 0.5% Xylocaine with 6 mg of non-particulate Celestone.
  Interventions: Drug: Xylocaine; Drug: Xylocaine and Celestone

INTERVENTIONS:
Drug: Xylocaine — 0.5% Xylocaine
Drug: Xylocaine and Celestone — non-particulate Celestone
  Other Names: Celestone
  Arms: Xylocaine and Celestone

SUMMARY:
To study improvements or lack thereof with the interlaminar epidural patients with or without steroids experiences mid back, upper back or neck pain with or without chest wall and upper extremity pain of at least 6-months duration non-responsive to conservative management.

DETAILED DESCRIPTION:
This is a Single-center, prospective, controlled, double-blind, randomized study in thoracic and cervical regions.

Patients are studied in 2 groups in each region.

* Group I-local anesthetic only.
* Group II-local anesthetic with 6 mg of non-particulate Celestone.

All patients will be unblinded at 12 or 24 months. Non-responsive patients will be unblinded after 3 months and will be crossed over to a different group, if patient consents. Non-responsive patients may be unblinded and withdrawn from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of at least 18 years of age
* Subjects with a history of chronic, function-limiting thoracic or cervical pain with or without upper extremity pain of at least 6 months in duration
* Subjects who are able to give voluntary, written informed consent to participate in this investigation
* Subjects who, in the opinion of the PI, are able to understand this investigation, co-operate with the investigational procedures, and are willing to return to the center for all the required post-operative follow-ups
* Subjects have not had recent surgical procedures within the last 3 months.

Exclusion Criteria:

* Compressive radiculopathy
* Narcotic use of no greater than hydrocodone 100 mg/day, methadone of 60 mg, or morphine 180 mg, or dose equivalent
* Uncontrolled major depression or uncontrolled psychiatric disorders
* Uncontrolled or acute medical illnesses including coagulopathy, renal insufficiency, chronic liver dysfunction, progressive neurological deficit, urinary sphincter dysfunction, infection, increased intracranial pressure, pseudotumor cerebri, intracranial tumors, unstable angina, and severe chronic obstructive pulmonary disease
* Chronic severe conditions that could interfere with the interpretations of the outcome assessments for pain and bodily function
* Women who are pregnant or lactating
* Subjects who have participated in a clinical study with an investigational product within 30 days of enrollment
* Patients with multiple complaints involving concomitant shoulder osteoarthritis, due to the overlap of pain complaints
* Inability to achieve appropriate positioning and inability to understand informed consent and protocol
* History of adverse reaction to local anesthetic or anti-inflammatory drugs and history of gastrointestinal bleeding or ulcers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2008-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To demonstrate clinically significant improvements or lack thereof with the interlaminar epidural patients with or without steroids | Patients will return for follow-up visits at 3, 6, 12, 18, and 24 months post-treatment. The recruitment period is estimated as 24 months with an anticipated study duration of 48 months.
  examined improvements between those who received and did not receive steroids

SECONDARY OUTCOMES:
To evaluate differences in outcomes in patients receiving steroids compared to those patients randomized to the local anesthetic group who did not receive steroids. | Patients will return for follow-up visits at 3, 6, 12, 18, and 24 months post-treatment. The recruitment period is estimated as 24 months with an anticipated study duration of 48 months.
  examined differences between those who received and did not receive steroids
To evaluate and compare the adverse event profile in all patients. | Patients will return for follow-up visits at 3, 6, 12, 18, and 24 months post-treatment. The recruitment period is estimated as 24 months with an anticipated study duration of 48 months.
  examined adverse event differences between those who received and did not receive steroids

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, MD, Principal Investigator — Ambulatory Surgery Center, Paducah
Locations (1):
- Ambulatory Surgery Center, Paducah, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manchikanti L, Cash KA, Pampati V, Wargo BW, Malla Y. A randomized, double-blind, active control trial of fluoroscopic cervical interlaminar epidural injections in chronic pain of cervical disc herniation: results of a 2-year follow-up. Pain Physician. 2013 Sep-Oct;16(5):465-78. PMID 24077193
- [Derived] Manchikanti L, Malla Y, Cash KA, McManus CD, Pampati V. Fluoroscopic epidural injections in cervical spinal stenosis: preliminary results of a randomized, double-blind, active control trial. Pain Physician. 2012 Jan-Feb;15(1):E59-70. PMID 22270749
- [Derived] Manchikanti L, Malla Y, Cash KA, McManus CD, Pampati V. Fluoroscopic cervical interlaminar epidural injections in managing chronic pain of cervical postsurgery syndrome: preliminary results of a randomized, double-blind, active control trial. Pain Physician. 2012 Jan-Feb;15(1):13-25. PMID 22270734
- [Derived] Manchikanti L, Cash KA, McManus CD, Pampati V, Benyamin RM. A preliminary report of a randomized double-blind, active controlled trial of fluoroscopic thoracic interlaminar epidural injections in managing chronic thoracic pain. Pain Physician. 2010 Nov-Dec;13(6):E357-69. PMID 21102973
- [Derived] Manchikanti L, Cash KA, Pampati V, Wargo BW, Malla Y. Cervical epidural injections in chronic discogenic neck pain without disc herniation or radiculitis: preliminary results of a randomized, double-blind, controlled trial. Pain Physician. 2010 Jul-Aug;13(4):E265-78. PMID 20648213
- [Derived] Manchikanti L, Cash KA, Pampati V, Wargo BW, Malla Y. The effectiveness of fluoroscopic cervical interlaminar epidural injections in managing chronic cervical disc herniation and radiculitis: preliminary results of a randomized, double-blind, controlled trial. Pain Physician. 2010 May-Jun;13(3):223-36. PMID 20495586
- Available data/document: Clinical Study Report — http://painphysicianjournal.com/current/pdf?article=MTk3Nw%3D%3D&journal=77 — A Randomized, Double-Blind, Active Control Trial of Fluoroscopic Cervical Interlaminar Epidural Injections in Chronic Pain of Cervical Disc Herniation: Results of a 2-Year Follow-Up